CLINICAL TRIAL: NCT04412148
Title: Modified SALT Score for Assessment of Alopecia Areata
Brief Title: Modified SALT Score for Alopecia Areata
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: EgymSALT
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralesional Steroids (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide
- Control (Placebo Comparator)
  Interventions: Other: saline

INTERVENTIONS:
Drug: Triamcinolone Acetonide — intralesional injection of triamcinolone acetonide every 2 weeks for 6 sessions
  Arms: Intralesional Steroids
Other: saline — intralesional injection of saline
  Arms: Control

SUMMARY:
Patchy Alopecia areata was treated by intralesional steroids for 3 months and was evaluated by percentage of involvement, mSALT score and dermoscopy.

ELIGIBILITY:
Inclusion Criteria:

* localized scalp AA ( 2 patches and ≤50% scalp involvement , duration more than 6 months) • patients who did not receive any medication for at least 2 months before starting the study and those who agreed to join the study and signed written consent.

Exclusion Criteria:

* • pregnant, and lactating females

  * Alopecia totalis or universalis or ophiasis or cicatritial alopecia
  * Usage of systemic treatment of alopecia areata 2 months prior to the study.
  * Any scalp lesion within the treated area
  * Bleeding diathesis, severe anemia or platelet disorders
  * Medical conditions such as autoimmune diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage involvement | 6months to 1 year
  Degree of severity expressed as a percentage
Modified Severity of Alopecia Tool (mSALT) score | 6 months to 1 year
  New Score calculating severity (hair density) and area as a number minimum value is 0 and maximum value is 105 the higher the number of the score the worse the affection

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy university hospital, Faulty of medicine,Cairo university, Cairo, Egypt